CLINICAL TRIAL: NCT02966327
Title: Effect of Early Compression Therapy and Individualized Exercise on Incidence of Lymphedema in Patients Treated for Gynecological Cancer: a Pilot Randomized Controlled Trial
Brief Title: Effect of Early Compression and Exercise on Lymphedema Incidence in Patients With Gynecological Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Shirin M. Shallwani, Physiotherapist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A11-M104-14B
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Genital Neoplasms, Female; Lymphedema
MeSH Terms: conditions — Genital Neoplasms, Female; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compression Stockings-Exercise (Experimental): At T2 (4-6 weeks post-operatively), 25 study participants will be randomized to the intervention group and will be prescribed compression stockings and individualized exercise. They will also receive standard education on lymphedema risk reduction.
  Interventions: Device: Bilateral leg compression stockings; Behavioral: Individualized exercise; Behavioral: Lymphedema risk reduction
- Control Group (Other): At T2 (4-6 weeks post-operatively), 25 study participants will be randomized to the control group and will receive standard education on lymphedema risk reduction.
  Interventions: Behavioral: Lymphedema risk reduction

INTERVENTIONS:
Device: Bilateral leg compression stockings — Prescribed Jobst Elvarex compression class 1 (18 to 21 mmHg) standard or custom-made stockings for both lower limbs with or without panty; participants will be recommended to wear the garments for 12 to 16 hours daily for at least 6 months post-operatively.
  Arms: Compression Stockings-Exercise
Behavioral: Individualized exercise — Individualized education on exercise according to the Canadian Physical Activity Guidelines and self-lymphatic drainage techniques
  Arms: Compression Stockings-Exercise
Behavioral: Lymphedema risk reduction — Standard education on lymphedema risk reduction along with printed materials from the Lymphedema Association of Quebec

SUMMARY:
Objectives: 1) To evaluate the effect of early compression therapy with individualized exercise on the incidence of lower limb lymphedema at 12 months post-operatively in patients treated for gynecological cancer who are at risk of developing lymphedema; 2) To evaluate the effect of early compression therapy with individualized exercise on lower limb volume, quality of life and incidence of cellulitis infections at 12 months post-operatively in this population.

DETAILED DESCRIPTION:
Study design and setting: A pilot randomized controlled trial will be conducted on 50 patients with gynecological cancer recruited from the McGill University Health Centre (MUHC) Royal Victoria Hospital and the Jewish General Hospital (JGH) Segal Cancer Centre in Montreal, Quebec. The data collection and interventions will be conducted at the MUHC Lymphedema Support Centre.

Intervention: At 4-6 weeks post-operatively, each participant in the experimental group will be prescribed Jobst Elvarex compression class 1 (18 to 21 mmHg) standard or custom-made stockings for both lower limbs with or without panty. The participants will be recommended to wear the garments for 12 to 16 hours daily for at least 6 months post-operatively. At this time, the participants will also receive individualized education on exercise, self-lymphatic drainage and skin care by an unblinded lymphedema therapist.

Control: At 4-6 weeks post-operatively (T2), both groups will receive standard education on lymphedema risk reduction along with printed materials from the Lymphedema Association of Quebec.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age;
* diagnosis of grade 2 or 3 endometrial cancer, or high grade type (serous or clear cell), stage 1b1 or stage 2a cervical cancer, stage 1 vulvar cancer with tumor greater than 4 cm, or stage 2 or 3 vulvar cancer;
* to undergo surgical lymph node dissection.

Exclusion Criteria:

* recurrent diagnosis of gynecological cancer;
* presence of distant metastases (stage 4 cancer);
* body mass index of 35 or greater.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in bilateral lower limb volume | Prior to surgery (T1), at 4-6 weeks post- operatively (T2), at 3 months post-operatively (T3), at 6 months post-operatively (T4) and at 1 year post-operatively (T5)
  Measured with circumferential measures and perometry (Perometer 350S)

SECONDARY OUTCOMES:
Change in bilateral lower limb extracellular fluid volume | Prior to surgery (T1), at 4-6 weeks post- operatively (T2), at 3 months post-operatively (T3), at 6 months post-operatively (T4) and at 1 year post-operatively (T5)
  Measured with bioimpedance spectroscopy
EORTC QLQ-C30 questionnaire | Prior to surgery (T1), at 4-6 weeks post- operatively (T2), at 3 months post-operatively (T3), at 6 months post-operatively (T4) and at 1 year post-operatively (T5)
  Measure of quality of life
Incidence of cellulitis | Prior to surgery (T1), at 4-6 weeks post- operatively (T2), at 3 months post-operatively (T3), at 6 months post-operatively (T4) and at 1 year post-operatively (T5)
  Patient-reported number of cellulitis infections

CONTACTS AND LOCATIONS:
Overall Officials: Shirin M. Shallwani, MSc, PT, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Anna Towers, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre Lymphedema Support Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shallwani SM, Towers A, Newman A, Salvador S, Yung A, Gilbert L, Gotlieb WH, Zeng X, Thomas D. Feasibility of a Pilot Randomized Controlled Trial Examining a Multidimensional Intervention in Women with Gynecological Cancer at Risk of Lymphedema. Curr Oncol. 2021 Jan 13;28(1):455-470. doi: 10.3390/curroncol28010048. PMID 33450972